CLINICAL TRIAL: NCT07271927
Title: Evaluation Study of the Effects and Safety of Whole-Body Photobiomodulation Therapy on Motor and Cognitive Changes in Patients With Parkinson's Disease
Brief Title: Whole-Body Photobiomodulation for Motor and Cognitive Changes in Parkinson's Disease
Acronym: PBM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Professor, Pusan National University Yangsan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-2024-005
Record Dates: First submitted 2025-08-21; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: Photobiomodulation; Parkinson disease; cognition; motor function; light theraphy
MeSH Terms: conditions — Parkinson Disease | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parkinson (Experimental): Participants received whole-body PBM therapy once daily (20 minutes per session), three times per week, for approximately 10 weeks, totaling 30 sessions.
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — Participants received whole-body PBM therapy over approximately 10 weeks (three sessions per week, once daily, 20 minutes per session), with each session using a randomly selected wavelength of either 660 nm, 850 nm, or 940 nm (±20%).

SUMMARY:
This study aims to exploratorily evaluate the extent of motor and cognitive changes, as well as the safety, resulting from approximately 10 weeks of whole-body photobiomodulation (PBM) therapy (about three sessions per week, once daily, 20 minutes per session) in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with Parkinson's disease at Hoehn and Yahr stages 1-3 based on medical history and examination
* Adults aged 40 years or older
* Individuals able to walk independently

Exclusion Criteria:

* Individuals with severe cognitive impairment (Korean Mini-Mental State Examination [K-MMSE] score ≤ 9) making it difficult to understand and perform tasks
* Patients with dementia other than Parkinson's disease dementia
* Individuals with implanted medical or other electronic devices
* Individuals with severe neuropsychiatric disorders
* Individuals treated for alcohol dependence within 6 months prior to screening
* Individuals with a history of suicide attempts
* Individuals with a history of seizures
* Individuals experiencing dyspnea while sitting at rest
* Individuals with visual impairment preventing them from reading ordinary text even with corrective lenses
* Individuals with hearing impairment preventing them from understanding conversation even with a hearing aid
* Individuals who have participated in two or more clinical trials in the same year or in another clinical trial within the past 6 months
* Women and men of childbearing potential who are planning pregnancy during the trial or who do not agree to use appropriate contraceptive methods
* Pregnant or breastfeeding women
* Individuals deemed medically inappropriate for participation by the principal investigator or study staff based on clinically significant findings not otherwise specified above

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
UPDRS | Change in UPDRS from baseline to post 30 sessions (up to approximately 10 weeks). The UPDRS ranges from 0 to 199, with higher scores indicating greater symptom severity.
  Unified Parkinson's Disease Rating Scale

SECONDARY OUTCOMES:
BBS | Change in Berg Balance Scale scores from baseline to post 30 sessions (up to approximately 10 weeks). The BBS ranges from 0 to 56, with higher scores indicating better balance performance.
  Berg Balance Scale
Grip strength and pinch strength test | Change in Grip strength and pinch strength from baseline to post 30 sessions (up to approximately 10 weeks). Higher scores indicate better hand function.
  Grasp, tip pinch & three jaw chuck
FRT | Change in Functional Reach Test scores from baseline to post 30 sessions (up to approximately 10 weeks). Higher scores indicate better hand function.
  Functional Reach Test
TUG | Change in Timed Up and Go test scores from baseline to post 30 sessions (up to approximately 10 weeks). Lower scores indicate better functional mobility.
  Timed Up and Go
CTRS | Change in CRTS scores from baseline to post 30 sessions (up to approximately 10 weeks). The score ranges from 0 to 160, with higher scores indicating more severe tremor symptoms.
  Clinical Rating Scale for Tremor
SVLT | Change in SVLT scores from baseline to post 30 sessions (up to approximately 10 weeks). The scores ranging from 0 to 36, where higher scores reflect better memory performance.
  Seoul verbal learning test
RCFT | Change in RCFT scores from baseline to post 30 sessions (up to approximately 10 weeks). Higher scores indicate better visuospatial and memory performance.
  Rey complex figure test
DST | Change in DST scores from baseline to post 30 sessions (up to approximately 10 weeks). Higher scores indicate better performance.
  Digit span test
TMT | Change in TMT scores from baseline to post 30 sessions (up to approximately 10 weeks). Faster completion times (i.e., lower scores) indicate better cognitive function.
  Trail making test
K-CWST | Change in K-CWST scores from baseline to post 30 sessions (up to approximately 10 weeks). Faster completion times (i.e., lower scores) indicate better cognitive function.
  Korean-Color word stroop test

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) cannot be shared due to protection of participants' personal information and regulatory restrictions of our hospital.